CLINICAL TRIAL: NCT05179226
Title: A Phase III, Prospective, Open-label, Multi-center Trial of Ferric Derisomaltose in Children 0 to <18 Years of Age With Iron Deficiency Anemia Due to NDD-CKD or With Iron Deficiency Anemia Who Are Intolerant or Unresponsive to Oral Iron
Brief Title: Multi-center Trial of Ferric Derisomaltose in Children 0 to <18 Years of Age With Iron Deficiency Anemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-PED-01; U1111-1266-9073 (Registry Identifier: WHO)
Record Dates: First submitted 2021-11-16; First posted 2022-01-05 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency, Anaemia in Children
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric derisomaltose

STUDY DESIGN:
Intervention Model Description: The study includes a PK-part. 24 subjects will be part of a PK assessment and have total- iron PK-parameters measured 7 or 8 times between baseline visit and week 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferric Derisomaltose (Experimental): All subjects (a total of 200) will be treated with Ferric Derisomaltose. 12 subjects (half of the 24 subjects participating in the PK-part of the trial) will be treated with 10mg/kg while the remaining subjects will be treated with 20 mg/kg.
  .
  Interventions: Drug: Ferric Derisomaltose

INTERVENTIONS:
Drug: Ferric Derisomaltose — All subjects will be treated with Ferric derisomaltose 20 mg/kg at baseline visit except for 12 subjects included in the PK-group, who will be treated with 10 mg/kg
  Other Names: Monofer®, Monoferric®

SUMMARY:
Several clinical trials have been reported for ferric derisomaltose where it has been shown to be well tolerated and to improve markers of IDA. All clinical trials with ferric derisomaltose have been performed in adults, however, IDA is not specific to the adult population. In fact, children are likely to develop IDA due to their rapid growth.

The aim in this trial is to evaluate the efficacy and safety of intravenous (IV) ferric derisomaltose in children 0 to <18 years of age with IDA due to NDD-CKD or with IDA who are intolerant or unresponsive to oral iron .

The subjects will receive ferric derisomaltose/iron isomaltoside 1000 (Monoferric®/Monofer®), at single doses of 10 mg/kg or 20 mg/kg with a maximal dose of 1000 mg.

24 subjects will be part of a PK assessment, meaning that more blood samples will be drawn within the first week after treatment. The blood samples will be used for analysis of the amount of total iron in the blood from treatment is given to day 7.

For the individual subject, duration of the trial will be approximately 10 weeks (including a 14-day screening period) and each subject will attend 6-9 visits. Subjects who will be included in the PK assessments will attend 8 (subjects age 6 to <12 years old and 0 to <6 years old) or 9 (subjects age 12 to <18 years old) visits, while the other subjects will attend 6 visits.

DETAILED DESCRIPTION:
This is a combined clinical pharmacology and phase III study. The study is a prospective, open-label, multi-center study. Children 0 to <18 years of age with iron deficiency anemia (IDA) with a) non-dialysis dependent chronic kidney disease (NDD-CKD) or b) who are intolerant or unresponsive to oral iron will be enrolled. The subjects will receive ferric derisomaltose/iron isomaltoside 1000 (Monoferric®) at single doses of 10 mg/kg or 20 mg/kg with a maximal dose of 1000 mg.

A total of 200 subjects will be enrolled. Of these will 24 be part of the PK assessment. PK-subjects will be included in cohorts of 4 with the oldest age group as the first and with ferric derisomaltose 10 mg/kg to be increased to 20 mg/kg for the next cohort. Thus 12 subjects will be treated with 10mg/kg and the remaining 188 subjects with 20mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects <18 years
* Informed consent and child assent, as age-appropriate, obtained before any trial- related activities and willingness to participate. LAR of the subject must sign and date the ICF (according to local requirements). The child must sign and date the CAF or provide oral assent, if required according to local requirements
* IDA caused by different etiologies such as gastrointestinal disease, NDD-CKD, or other conditions leading to IDA
* Hb concentration less than the 5th percentile for age and sex-specific reference range (Appendix B)
* Subjects with NDD-CKD (a) or who are intolerant or unresponsive to oral iron (b):

  a) Subjects with NDD-CKD:
* TSAT ≤35 % or s-ferritin <100 ng/mL
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2
* If on ESA, receiving stable ESA regimen defined as dose adjustments no more than

  ± 20 % for ≥8 weeks prior to screening

  b) Subjects with documented history of intolerance or unresponsiveness to oral iron therapy for at least one month prior to trial enrolment.
* TSAT ≤20 % or s-ferritin <100 ng/mL

Exclusion Criteria:

* Anemia caused by factors other than IDA according to Investigator's judgment
* S-ferritin >600 ng/mL
* Hb ≤5.0 g/dL
* Iron overload or disturbances in utilization of iron (e.g. hemochromatosis and hemosiderosis)
* ALAT and/or ASAT >2 times upper limit of normal (e.g. decompensated liver cirrhosis or active hepatitis)
* Pregnant or nursing female subjects. In order to avoid pregnancy, female subjects of childbearing potential have to use adequate contraception (e.g. intrauterine devices, hormonal contraceptives, or double barrier method) or be abstinent during the whole trial period and 7 days after the last dosing. Childbearing potential refers to all female subjects ≥12 years old or <12 years old who have started menstruating
* Previous serious hypersensitivity reactions to any IV iron compounds including ferric derisomaltose
* Received an investigational drug within 30 days prior to screening
* Treatment with IV iron within 10 days prior to screening
* Treatment with blood transfusion, radiotherapy, chemotherapy or other drugs that suppress the bone marrow, and drugs which have anemia as side effect within 30 days prior to screening
* Planned elective surgery (or planned surgery during the trial period) where significant blood loss is expected within the last 30 days prior to screening
* Any non-viral infection (non-viral infection that has been fully treated before the baseline visit is accepted)
* Any other laboratory abnormality, medical condition, or psychiatric disorders which, in the opinion of the Investigator, will put the subject's disease management at risk or may result in the subject being unable to comply with the trial requirements

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of subjects with a Hb increase of ≥1 g/dL (NDD-CKD) or 2 g/dL (intolerant or unresponsive to oral iron). Measurement by bloodsample. | From baseline at any time from week 1 to week 8
  Hb (g/dL), measurement by bloodsample analysis

SECONDARY OUTCOMES:
Time to increase Hb ≥1 g/dL (NDD-CKD) or 2 g/dL (intolerant or unresponsive to oral iron). Measurement by bloodsample. | From baseline at any time from week 1 to week 8
  Hb (g/dL), measurement by bloodsample analysis
Incidence of subjects who achieve a serum (s-) ferritin of ≥100 ng/mL. Measurement by bloodsample. | At weeks 1, 2, 4, and 8
  s-ferritin (ng/mL), measurement by bloodsample analysis
Incidence of subjects who achieve a TSAT of ≥35 % (NDD-CKD) or ≥20 % (intolerant or unresponsive to oral iron). Measurement by bloodsample. | At weeks 1, 2, 4, and 8
  TSAT (%), measurement by bloodsample analysis
Total iron PK parameters: AUC0-∞ | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Total iron PK parameters: AUC0-t | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Total iron PK parameters: Cmax | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Total iron PK parameters: Tmax | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Total iron PK parameters: Ke | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Total iron PK parameters: T½ | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Total iron PK parameters: CL | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Total iron PK parameters: Vd | From baseline to day 7
  Total iron (µg/dL), measurement by bloodsample analysis
Type and incidence of AEs | From baseline to week 8
  Any AE
Serious or severe hypersensitivity reaction | From treatment (Baseline) to 24 hours
  Any serious or severe hypersensitivity reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacosmos Investigational Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No